CLINICAL TRIAL: NCT06225037
Title: EEG-guided Propofol Sedation Versus Standard Care for Oesophagogastroduodenoscopy and Colonoscopy in Children: A Randomised Controlled Trial to Improve Sedation Safety and Experience
Brief Title: EEG-guided Propofol Sedation Versus Standard Care for Oesophagogastroduodenoscopy and Colonoscopy in Children
Acronym: EPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/2337
Record Dates: First submitted 2023-12-19; First posted 2024-01-25 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Anesthesia; Adverse Effect; Anesthesia Emergence Delirium; Sedation Complication; Sedative Adverse Reaction
Keywords: EEG-guided sedation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: EEG Monitoring (Experimental): EEG sensor placed with the EEG monitored.
  Interventions: Device: Sedline EEG monitoring
- Group 2: Standard Care (Active Comparator): EEG sensor placed with the output concealed.
  Interventions: Device: Sedline EEG with output concealed

INTERVENTIONS:
Device: Sedline EEG monitoring — Propofol titrated according to the raw EEG and spectrogram, aiming to maintain sedation (alpha oscillations +/- slow oscillations) and preventing burst suppression, keeping the PSI greater than 25 where possible.
  Arms: Group 1: EEG Monitoring
Device: Sedline EEG with output concealed — Clinician will be blinded to the sedline output but data will be collected for analysis (Sedline output will only be analysed at data analysis)
  Arms: Group 2: Standard Care

SUMMARY:
The goal of this clinical trial is to compare electroencephalogram (EEG) guided propofol sedation versus standard care in paediatric patients aged 6-16 undergoing oesophagogastroduodenoscopy and colonoscopy. The main questions it aims to answer are whether EEG guided propofol sedation will result in:

* faster wake up time
* reduced time to discharge
* reduced cumulative propofol dosage
* lower incidence of intraoperative adverse events
* no difference in intraoperative undesirable movement
* lower incidence and severity of emergence delirium
* lower intraoperative depth of sedation Participants will wear an EEG sensor (Sedline) prior to undergoing propofol sedation until they wake up post procedure.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Oesophagogastroduodenoscopy (OGD) and colonoscopy in children are often performed under deep sedation with propofol. Titration of propofol dosage is based solely on cardiorespiratory parameters obtained from standard ASA monitoring. However, this method of propofol titration does not allow visualisation of the patients' brain response and often leads to under- or over-sedation. Under-sedation can lead to undesirable intra-operative movement and potential awareness, while over-sedation is associated with complications such as apnea, hypoxaemia, hypotension, prolonged time to awakening and delay in PACU discharge.(1,2)

Patients are often over-sedated during propofol anaesthesia. A study in adults undergoing colonoscopy using electroencephalography (EEG) monitoring showed that although providers planned for moderate-to-deep sedation, retrospective review of the EEG revealed that many patients were under general anesthesia, often with burst suppression (3) EEG burst suppression has been linked to postoperative deliriumin the elderly (4), and anesthesia titration to minimize burst suppression may decrease the incidence of postoperative delirium. Likewise, over-sedation and EEG isoelectric events are common in children undergoing propofol anesthesia with dosing based solely on population pharmacokinetics and patient haemodynamics. (5)

It was recently proposed that EEG monitoring and guidance during anaesthesia and sedation in children allows direct visualisation of each patient's brain response and complements current standard monitoring to enhance patient safety and experience.(2) EEG-guidance has been shown to reduce sevoflurane requirements in children undergoing general anaesthesia. (9) In particular, the EEG spectrogram, also called density spectral array (DSA), allows easy visualisation of the interactions between brain response, hemodynamic response, and changing procedural stimulation in real time, thus facilitating more precise and nuanced titration of anaesthetic agents. (2)

Processed EEG (pEEG) such as the bispectral index (BIS), Narcotrend index (NI) and patient state index (PSI) are dimensionless numbers derived from the EEG using manufacturers' algorithms to quantify anaesthetic depth (6). However, given the lack of clarity on how different pEEG numbers are computed and how they relate to fundamental neurophysiological properties of the developing brain, it is important to interpret the pEEG number in relation to the raw EEG waveform and spectrogram.

Only two small studies have compared EEG-guided propofol anaesthesia with standard care in children, both using the Narcotrend Index (NI). NI-guidance was shown to result in slightly faster recovery and lower drug consumption.(7)(8). To date, no study has utilised the spectrogram together with the pEEG number to guide anaesthesia. The investigators aim to compare EEG-guidance using Sedline EEG and spectrogram, in addition to the PSI, with standard care in children undergoing propofol TIVA for OGD and colonoscopy. Better visualisation of the brain response using the spectrogram may lead to more precise titration of propofol doses, lower propofol consumption and greater reduction in wake up time.

List of references:

1. Patino M, Glynn S, Soberano M, Putnam P, Hossain MM, Hoffmann C, Samuels P, Kibelbek MJ, Gunter J. Comparison of different anesthesia techniques during esophagogastroduedenoscopy in children: a randomized trial. Paediatr Anaesth. 2015;25:1013-1019. Cited: in: : PMID: 26184697.
2. Bong CL, Balanza GA, Khoo CE-H, Tan JS-K, Desel T, Purdon PL. A Narrative Review Illustrating the Clinical Utility of Electroencephalogram-Guided Anesthesia Care in Children. Anesth Analg [Internet]. 2022; doi: 10.1213/ANE.0000000000006267. Cited: in: : PMID: 36729437.
3. Bloom J, Wyler D, Torjman MC, Trinh T, Li L, Mehta A, Fitchett E, Kastenberg D, Mahla M, Romo V. High Incidence of Burst Suppression during Propofol Sedation for Outpatient Colonoscopy: Lessons Learned from Neuromonitoring. Anesthesiol Res Pract. 2020;2020:7246570. Cited: in: : PMID: 32636880.
4. Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016;122:234-242. Cited: in: : PMID: 26418126.
5. Yuan I, Landis WP, Topjian AA, Abend NS, Lang S-S, Huh JW, Kirschen MP, Mensinger JL, Zhang B, Kurth CD. Prevalence of Isoelectric Electroencephalography Events in Infants and Young Children Undergoing General Anesthesia. Anesth Analg. 2020;130:462-471. Cited: in: : PMID: 31107263.
6. Soehle M, Kuech M, Grube M, Wirz S, Kreuer S, Hoeft A, Bruhn J, Ellerkmann RK. Patient state index vs bispectral index as measures of the electroencephalographic effects of propofol. Br J Anaesth. 2010;105:172-178. Cited: in: : PMID: 20587537.
7. Weber F, Walhout LC, Escher JC. The impact of NarcotrendTM EEG-guided propofol administration on the speed of recovery from pediatric procedural sedation-A randomized controlled trial. Paediatr Anaesth. 2018;28:443-449. Cited: in: : PMID: 29575232.
8. Weber F, Pohl F, Hollnberger H, Taeger K. Impact of the Narcotrend Index on propofol consumption and emergence times during total intravenous anaesthesia with propofol and remifentanil in children: a clinical utility study. Eur J Anaesthesiol. 2005;22:741-747. Cited: in: : PMID: 16211731.
9. Long MHY, Lim EHL, Balanza GA, Allen JC Jr, Purdon PL, Bong CL. Sevoflurane requirements during electroencephalogram (EEG)-guided vs standard anesthesia Care in Children: A randomized controlled trial. J Clin Anesth. 2022;81:110913. Cited: in: : PMID: 35772250.

HYPOTHESIS AND OBJECTIVES The primary hypothesis is that in children aged 6-16, personalised EEG-guided anaesthesia care using the Sedline, (based on the raw EEG, density spectral array, in addition to the patient state index (PSI)), will result in faster wake up (defined as time from end of procedure to time of first eye opening) after propofol sedation for OGD and colonoscopy by 8 minutes.

Our secondary hypotheses are that in children aged 6 to 16, personalised EEG-guided anaesthesia care using the Masimo Sedline, (based on the unprocessed EEG, density spectral array, in addition to the patient state index (PSI)) leads to:

1. A reduction in time to discharge from PACU (defined as time from PACU arrival to time of meeting PACU discharge criteria) by 15 minutes
2. A reduction of propofol dosage (cumulative/kg/time) by 10%
3. Lower incidence of intraoperative adverse events: apnea, hypoventilation requiring bag mask ventilation, laryngospasm, hypotension.
4. No difference in intraoperative undesirable movement
5. Lower Incidence and severity of emergence delirium as measured by the Paediatric Anaesthesia Emergence Delirium (PAED) scale
6. Lower intra-operative depth of sedation as measured by incidence and duration of burst suppression, intra-operative spectral edge frequency; alpha power and frequency; slow power and frequency.

Our primary aim is to determine if personalised EEG-guided anaesthesia care using the Sedline reduces the time to wake up after propofol sedation for oesophagogastroduodenoscopy (OGD) and colonoscopy.

Our secondary aims are to determine if personalised EEG-guided anaesthesia care reduces

1. Time to discharge from PACU
2. Total propofol dose used (cumulative mg/kg/min)
3. Incidence of intraoperative adverse events: apnea, hypoventilation requiring bag mask ventilation, laryngospasm, hypotension
4. Incidence of intra-operative undesirable movement
5. Incidence and severity of emergence delirium
6. Intra-operative depth of sedation

Inclusion Criteria

Subjects must meet all of the inclusion criteria to participate in this study. Inclusion Criteria:

1. Paediatric patients aged 6-16 who are undergoing oesophagogastroduodenoscopy and colonoscopy in KKH under propofol sedation
2. Parent/guardian must consent to participation in the study and patient must assent to participation in the study

Exclusion Criteria

Subjects meeting any of the exclusion criteria at baseline will be excluded from participation in the study. Exclusion Criteria:

1. Patients with neurological diseases including seizure disorders
2. Patients with developmental delay or genetic syndromes
3. Patients with craniofacial deformities where it is not possible to place the EEG sensors
4. Patients with severe eczema or skin allergy or atopy
5. Patients who require sedative premedication or who require inhalational induction prior to initiation of propofol sedation

STUDY DESIGN AND PROCEDURES/METHODOLOGY This is a single centre randomized controlled study of 50 children aged 6-16 years of age undergoing oesophagogastroduodenoscopy or colonoscopy under intravenous anaesthesia with propofol.

Following institutional ethics approval and written informed consent, children aged 6 to 16 receiving propofol sedation for colonoscopy lasting will be randomised in a 1:1 ratio to either:

Group 1: EEG Monitoring: EEG sensor placed with the EEG monitored. Propofol titrated according to the raw EEG and spectrogram, aiming to maintain sedation (alpha oscillations +/- slow oscillations) and preventing burst suppression, keeping the PSI greater than 25 where possible.

Group 2: Standard Care: EEG sensor placed with the output concealed. The anaesthesia team is blinded to the EEG data. Propofol is titrated according to routine standard care.

The EEG sensor will be placed over the forehead prior to induction of anaesthesia, and removed once the patient is awake at the conclusion of general anaesthesia. Routine monitors including ECG, pulse oximetry and non-invasive blood pressure will be placed and the patients managed according to standard care.

The pharynx will be tropicalized with 10% Xylocaine spray prior to insertion of the endoscope.

Fentanyl 0.5 mcg/kg and lignocaine 0.5mg/kg will be given prior to induction.

Propofol target controlled infusion (TCI) - Paedfusor model, will be used. The induction dose will be Cp 4.0mcg/ml and then titrated to patient response with (group 1) or without (group 2) EEG guidance.

Intra-operatively, the details of the anaesthetic, including the duration of sedation, TCI dosage at different pre-specified time points and cumulative propofol dosage, will be recorded. EEG characteristics during insertion of scope, maintenance, removal of scope and emergence will be noted. Any undesirable intraoperative patient movements, adverse events including apnea, hypoventilation requiring bag mask ventilation, laryngospasm, hypotension will also be recorded.

In the PACU, the time to wake up, time to PACU discharge, and the incidence and severity of emergence delirium will be recorded. The EEG information will be downloaded and anonymised for analysis. The incidence and duration of burst suppression, spectral edge frequency; alpha power and frequency; slow power and frequency will be recorded.

The investigators will compare the:

1. Time to wake up (defined as time from end of procedure to time of first eye opening)
2. Time to discharge from PACU (defined as time from PACU arrival to time of meeting PACU discharge criteria)
3. Total propofol dose used (cumulative mg/kg/min)
4. Incidence of intraoperative adverse events: apnea, hypoventilation requiring bag mask ventilation, laryngospasm, hypotension
5. Incidence of intra-operative undesirable movement
6. Incidence and severity of emergence delirium (as measured by the Paediatric Anaesthesia Emergence Delirium (PAED) scale)
7. Intra-operative depth of sedation (as measured by incidence and duration of burst suppression, intra-operative spectral edge frequency; alpha power and frequency; slow power and frequency)

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric patients aged 6-16 who are undergoing oesophagogastroduodenoscopy and colonoscopy in KKH under propofol sedation
2. Parent/guardian must consent to participation in the study and patient must assent to participation in the study

Exclusion Criteria:

1. Patients with neurological diseases including seizure disorders
2. Patients with developmental delay or genetic syndromes
3. Patients with craniofacial deformities where it is not possible to place the EEG sensors
4. Patients with severe eczema or skin allergy or atopy
5. Patients who require sedative premedication or who require inhalational induction prior to initiation of propofol sedation

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Time to wake up | Through study completion, approximately 6 months
  Our primary hypothesis is that in children aged 6-16, personalised EEG-guided anaesthesia care using the Sedline, (based on the raw EEG, density spectral array, in addition to the patient state index (PSI)), will result in faster wake up (defined as time from end of procedure to time of first eye opening) after propofol sedation for OGD and colonoscopy by 8 minutes

SECONDARY OUTCOMES:
Time to discharge | Through study completion, approximately 6 months
  A reduction in time to discharge from PACU (defined as time from PACU arrival to time of meeting PACU discharge criteria) by 15 minutes
Propofol dosage | Through study completion, approximately 6 months
  A reduction of propofol dosage (cumulative/kg/time) by 10%
Intraoperative adverse events | Through study completion, approximately 6 months
  Lower incidence of intraoperative adverse events: apnea, hypoventilation requiring bag mask ventilation, laryngospasm, hypotension.
Undesirable movement | Through study completion, approximately 6 months
  No difference in intraoperative undesirable movement
Emergence delirium | Through study completion, approximately 6 months
  Lower Incidence and severity of emergence delirium as measured by the "Paediatric Anaesthesia Emergence Delirium scale" (PAED scale), a scale from 0-20 where higher scores indicate a worse outcome.
Depth of sedation | Through study completion, approximately 6 months
  Lower intra-operative depth of sedation as measured by incidence and duration of burst suppression, intra-operative spectral edge frequency; alpha power and frequency; slow power and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Choon Looi Bong, Principal Investigator — Singhealth Foundation
Locations (1):
- KK Women and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patino M, Glynn S, Soberano M, Putnam P, Hossain MM, Hoffmann C, Samuels P, Kibelbek MJ, Gunter J. Comparison of different anesthesia techniques during esophagogastroduedenoscopy in children: a randomized trial. Paediatr Anaesth. 2015 Oct;25(10):1013-9. doi: 10.1111/pan.12717. Epub 2015 Jul 17. PMID 26184697
- [Background] Bong CL, Balanza GA, Khoo CE, Tan JS, Desel T, Purdon PL. A Narrative Review Illustrating the Clinical Utility of Electroencephalogram-Guided Anesthesia Care in Children. Anesth Analg. 2023 Jul 1;137(1):108-123. doi: 10.1213/ANE.0000000000006267. Epub 2023 Jun 16. PMID 36729437
- [Background] Bloom J, Wyler D, Torjman MC, Trinh T, Li L, Mehta A, Fitchett E, Kastenberg D, Mahla M, Romo V. High Incidence of Burst Suppression during Propofol Sedation for Outpatient Colonoscopy: Lessons Learned from Neuromonitoring. Anesthesiol Res Pract. 2020 Jun 19;2020:7246570. doi: 10.1155/2020/7246570. eCollection 2020. PMID 32636880
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Yuan I, Landis WP, Topjian AA, Abend NS, Lang SS, Huh JW, Kirschen MP, Mensinger JL, Zhang B, Kurth CD. Prevalence of Isoelectric Electroencephalography Events in Infants and Young Children Undergoing General Anesthesia. Anesth Analg. 2020 Feb;130(2):462-471. doi: 10.1213/ANE.0000000000004221. PMID 31107263
- [Background] Soehle M, Kuech M, Grube M, Wirz S, Kreuer S, Hoeft A, Bruhn J, Ellerkmann RK. Patient state index vs bispectral index as measures of the electroencephalographic effects of propofol. Br J Anaesth. 2010 Aug;105(2):172-8. doi: 10.1093/bja/aeq155. Epub 2010 Jun 29. PMID 20587537
- [Background] Weber F, Walhout LC, Escher JC. The impact of Narcotrend EEG-guided propofol administration on the speed of recovery from pediatric procedural sedation-A randomized controlled trial. Paediatr Anaesth. 2018 May;28(5):443-449. doi: 10.1111/pan.13365. Epub 2018 Mar 25. PMID 29575232
- [Background] Weber F, Pohl F, Hollnberger H, Taeger K. Impact of the Narcotrend Index on propofol consumption and emergence times during total intravenous anaesthesia with propofol and remifentanil in children: a clinical utility study. Eur J Anaesthesiol. 2005 Oct;22(10):741-7. doi: 10.1017/s0265021505001237. PMID 16211731
- [Background] Long MHY, Lim EHL, Balanza GA, Allen JC Jr, Purdon PL, Bong CL. Sevoflurane requirements during electroencephalogram (EEG)-guided vs standard anesthesia Care in Children: A randomized controlled trial. J Clin Anesth. 2022 Oct;81:110913. doi: 10.1016/j.jclinane.2022.110913. Epub 2022 Jun 27. PMID 35772250